CLINICAL TRIAL: NCT02166788
Title: Inguinal or Ilio-inguinal Lymphadenectomy for Patients With Metastatic Melanoma to Groin Lymph Nodes and no Evidence of Pelvic Disease on PET/CT Scan - A Randomised Phase III Trial (EAGLE FM)
Brief Title: Evaluation of Groin Lymphadenectomy Extent For Metastatic Melanoma
Acronym: EAGLE FM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Cancer Council New South Wales (Other); Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01.12
Record Dates: First submitted 2014-06-15; First posted 2014-06-18 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Melanoma to the Groin Lymph Nodes
Keywords: metastatic melanoma; groin lymph nodes; surgery; lymphadenectomy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Inguinal Lymphadenectomy (Other): Inguinal Lymphadenectomy (IL) is removal of the easily accessible superficial groin lymph nodes (LNs) and has a median LN retrieval of 11 lymph nodes
  Interventions: Procedure: Inguinal Lymphadenectomy
- Arm 2: Ilio-inguinal Lymphadenectomy (Other): Ilio-inguinal Lymphadenectomy (I-IL) is the removal of the same superficial groin lymp nodes (LN) removed during an IL but also combined with the more surgically complex removal of the ipsilateral pelvic LN. About twice as many LN are removed with I-IL compared to IL.
  Interventions: Procedure: Ilio-inguinal Lymphadenectomy

INTERVENTIONS:
Procedure: Inguinal Lymphadenectomy
  Arms: Arm 1: Inguinal Lymphadenectomy
Procedure: Ilio-inguinal Lymphadenectomy
  Arms: Arm 2: Ilio-inguinal Lymphadenectomy

SUMMARY:
BACKGROUND: Spread of metastatic melanoma to the groin lymph nodes (LN) is a common event affecting about 350 people a year in Australia. Globally it has been shown that patients with involved groin LN, without proven pelvic LN disease on imaging receive 1 of 3 management strategies in equal proportions - inguinal lymphadenectomy (IL); ilio-inguinal lymphadenectomy (I-IL); or variable use of either depending on circumstances. Different experts have strong and polarised opinions favouring either IL or more extensive I-IL with existing cases series reporting conflicting data on best cancer outcomes. No high level evidence proves which operation is best. HYPOTHESIS: There will be no significant difference in DFS between patients having IL or I-IL, conditional on PET/CT scan showing no evidence of pelvic disease at the time of diagnosis of groin LN metastatic melanoma. AIMS: To provide a rational evidence base for management for melanoma to the groin LNs by randomly assessing the effect of each operation on DFS, distant DFS, overall survival (OS), morbidity - including early complications and longer-term rates of lymphedema as well as comprehensively assessed QOL. Also to clarify the reliability of PET/CT scans for staging pelvic LNs and evaluate any health economic benefits of I-IL over IL. TARGET POPULATION: To recruit 634 patients in 5 years. DESIGN: An Australian led, international, multi-centre, non-inferiority, phase III, prospective, randomised clinical trial comparing IL or I-IL for patients with metastatic melanoma to groin LNs and no evidence of pelvic disease on PET/CT. ENDPOINTS: DFS, Distant DFS, OS and QOL at 5 years. Accuracy of PET/CT for pelvic LN metastases.

OUTCOMES: International standardization of care, improved cancer outcomes, improved QOL for patients with groin metastatic melanoma. Proof of principle about extent of surgery when PET/CT is clear in adjacent LN areas, leading to clinical trials investigating management of other lymph node fields.

DETAILED DESCRIPTION:
Background and Rationale

Spread of metastatic melanoma to the groin lymph nodes (LN) is a common event for patients with melanoma. In melanoma treatment centres around the world, patients without demonstrated pelvic LN disease receive 1 of 3 strategies of management in relatively equal proportions (Pasquali, Spillane et al. 2012):

i. Inguinal Lymphadenectomy (IL) ii. Ilio-inguinal Lymphadenectomy (I-IL) iii. Variable use of either IL or I-IL surgery.

Some larger melanoma centres have an institutional policy that all patients have either IL or I-IL for metastatic inguinal node involvement. Nearly all centres would agree that patients with pelvic LN involvement without distant metastatic disease should have I-IL.

Study Objectives This study aims to provide a more rational evidence base for appropriate management for metastatic melanoma in the groin LNs, through assessing the effect of the addition of ipsilateral pelvic lymphadenectomy on patient disease-free survival (DFS), distant disease-free survival (DDFS), overall survival (OS), morbidity, and quality of life. In addition, the study will clarify the reliability of PET (Positron Emission Tomography) / CT (Computed Tomography) scans for staging pelvic LNs, clarify morbidity differences between the operations in a balanced cohort, evaluate any health economic benefits of I-IL over IL and provide a tissue and serum resource to be used to identify biological markers of recurrence and progression after inguinal metastases.

Study Hypothesis There will be no significant difference in DFS between patients having IL or I-IL, conditional on PET/CT scan showing no evidence of pelvic disease at the time of diagnosis of groin LN metastatic melanoma.

Study Population The aim is to recruit 634 patients in 5 years who are 15 years or older with cytologically or histologically confirmed metastatic melanoma in inguinal LNs (H&E & IHC); specifically with no evidence of pelvic node involvement or distant spread of melanoma clinically or on PET/CT staging scans. To be eligible patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 at randomisation.

Study Treatments Eligible patients will be randomised 1:1 to undergo an IL or I-IL.

Study Design This is an international, multi-centre, phase III, non-inferiority, prospective, randomised clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

1. Must be 15 and above.
2. Have primary cutaneous melanoma or if the patient presents with stage III melanoma with no known primary tumour then a thorough search for the primary should be documented (including perineal and perianal areas)
3. Life expectancy of at least 10 years from the time of diagnosis, not considering the melanoma in question, as determined by the PI
4. Must have one or multiple inguinal node(s) involved, histologically or cytologically proven as metastatic melanoma. This can can be detected:

   * At the time of diagnosis;
   * Or by Ultrasound detection;
   * Or later after relapse when no Sentinel Node Biopsy (SNB) was performed at the time of primary tumour management;
   * Or as a result of SNB;
   * Or at the time of regional recurrence after "false negative" SNB;
5. Absent distant disease clinically and on PET/CT scan. (Patients must have NO further distant disease or visceral metastases)
6. ECOG performance status must be between 0 to 2 at randomisation
7. Whole body PET/CT scan, specifically stating there is NO evidence of pelvic lymph node involvement prior to randomisation and a CT Brain or MRI Brain scan. Scans must be performed within 6 weeks prior to randomisation.
8. Able to provide written, informed consent
9. Willing to return to the centre for follow up examinations and procedures, as outlined in the protocol.
10. All patients must be randomised and undergo lymphadenectomy surgery no more than 120 days following diagnosis of inguinal LN involvement

Exclusion Criteria:

1. Distant metastatic disease on clinical examination or staging imaging (CT/MRI brain or whole body PET/CT scan). Scans must be performed within 6 weeks prior to randomisation
2. Pelvic LN involvement on SNB or PET/CT scan suggestive of metastatic disease in the pelvis - criteria for diagnosis include normal size or enlarged lymph nodes (> 1 cm) with increased FDG activity on PET (SUV >3). If there are enlarged, necrotic lymph nodes FDG activity on PET is not required to be present. If unsure central review should be sought.
3. Bilateral inguinal lymph node involvement
4. Patients with a history of major pelvic surgery and / or regional radiotherapy at any time in the past
5. Requiring planned radiotherapy following surgery due to macroscopic, bulky and matted nodes.
6. Unfit for General Anaesthesia
7. Melanoma-related operative procedures not corresponding to criteria described in the protocol
8. Patients with prior cancers, except:

   * those with a thin <=1 mm, regionally unrelated melanoma > 5 years ago
   * those with a good prognosis regionally unrelated cancer (>90% probability of 10 years disease specific survival)
   * other cancers diagnosed more than five years ago with no evidence of disease recurrence within this time
   * successfully treated basal cell and squamous cell skin carcinoma
   * carcinoma in-situ of the cervix
   * 1 episode of in transit melanoma > 3 years ago
9. A medical or psychiatric condition that compromises ability to give informed consent or complete the protocol
10. Positive urine pregnancy test for women of childbearing potential (+/-7 days of randomisation onto the trial)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2015-03-02 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be Disease Free Survival following lymphadenectomy, assessed after 60 months of follow-up. | 60 Months
  The difference between IL and I-IL surgery in DFS 5 years after randomisation

SECONDARY OUTCOMES:
Overall Survival | 0 - 120 months
  time from randomisation to death from any cause
Distant Disease Free Survival | 0 - 120 Months
  time to new distant melanoma recurrence
Regional Recurrence Free Survival | 0 - 120 Months
  time to new regional lymph node recurrence
Morbidity differences | Up to 120 days from lymphadenectomy, and from 0 - 120 months
  This includes lymphoedema, wound complications (wound infections, dehiscence/necrosis, and seroma) chronic pain, and restriction in mobility
Quality Of Life | 0 - 120 Months
  Quality Of Life questionnaires completed by patients
Sensitivity / specificity and positive predictive value and negative predictive value of PET/CT for pelvic disease at diagnosis of groin LN involvement by melanoma. | 0 - 120 Months
  The diagnostic accuracy of PET/CT and CT for detecting pelvic lymph nodes positive for metastatic melanoma as confirmed by histopathology will be assessed in the sub-group of patients screened and shown to have a positive pelvic LN on PET/CT and those patients who had negative pelvic LN on PET/CT and randomised for I-IL treatment.
Resource use and utility based Quality Of Life | 0 - 60 Months
  Resource use will be identified from the trial case report forms, and valued according the relevant Australian Refined Diagnosis Related Groups and Medicare Benefits Schedule item numbers.The cost-effectiveness and cost-utility analyses will calculate total costs and mean per patient costs per surgical group allocation, as well as total and mean benefits per group allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spillane, Principal Investigator — The University of Sydney, Northern Clinical School
Locations (17):
- Australia (7):
  - Calvary Public Hospital Bruce, Canberra, Australian Capital Territory
  - Melanoma Institute Australia - The Poche Centre, North Sydney, New South Wales
  - Sydney Adventist Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Mater Hospital Brisbane, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Brazil (2):
  - Hospital de Câncer de Barretos, Barretos, São Paulo
  - A.C. Camargo Cancer Center, São Paulo, São Paulo
- Veneto Institute of Oncology - IOV, Padua, Veneto, Italy
- Netherlands (2):
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - University Medical Center Groningen, Groningen, Provincie Groningen
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- United Kingdom (4):
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Guy's and St Thomas's Hospitals, London
  - St George's Hospital, London
  - St Helen's and Knowsley Teaching Hospitals, St Helens

REFERENCES:
- [Derived] Mahumud RA, Law CK, Ospino DA, de Wilt JHW, van Leeuwen BL, Allan C, de Lima Vazquez V, Jones RP, Howle J, Peric B, Spillane AJ, Morton RL. Economic Evaluation of Inguinal Versus Ilio-inguinal Lymphadenectomy for Patients with Stage III Metastatic Melanoma to Groin Lymph Nodes: Evidence from the EAGLE FM Randomized Trial. Ann Surg Oncol. 2025 Jun;32(6):4211-4222. doi: 10.1245/s10434-025-17040-2. Epub 2025 Feb 27. PMID 40016616
- See also: Trial Website — https://www.masc.org.au/